CLINICAL TRIAL: NCT00490074
Title: A Phase I/II Trial to Compare the Immunogenicity and Safety of 3 DNA C Prime Followed by 1 NYVAC C Boost to 2 DNA C Prime Followed by 2 NYVAC C Boost
Brief Title: Study to Compare the Immunogenicity and Safety of Two HIV Preventive Vaccinations in Healthy Volunteers
Acronym: EV03/ANRSVAC20
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: EuroVacc Foundation (Other)
Responsible Party: Agence Nationale de la Recherche sur le Sida et les Hepatites virales (ANRS), French National Agency for Research on AIDS and Viral Hepatitis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2006-006141-13; EV03/ANRSVAC20
Record Dates: First submitted 2007-06-21; First posted 2007-06-22 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-11

CONDITIONS: HIV Infections
Keywords: AIDS Vaccines; Vaccines, DNA; HIV Preventive Vaccine; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — NYVAC-C vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3 DNA-C + 1 NYVAC-C (Experimental)
  Interventions: Biological: DNA-C; Biological: NYVAC-C
- 2 DNA-C + 2 NYVAC-C (Active Comparator)
  Interventions: Biological: DNA-C; Biological: NYVAC-C

INTERVENTIONS:
Biological: DNA-C — 1.0mg per ml of DNA HIV-C vaccine 2x2 ml IM
Biological: NYVAC-C — NYVAC-C 1 ml IM

SUMMARY:
The purpose of the trial is to evaluate the effect upon immune system of two regimens of preventive HIV vaccination in healthy adult volunteers. Volunteers will be vaccinated by DNA-C and NYVAC-C vaccines, and the immune changes will be assessed, as well as safety of the vaccines. Volunteers will be followed during 72 weeks.

DETAILED DESCRIPTION:
Methods: randomised phase I/II international trial with a parallel group design, open to participants and investigators but blind to laboratory personnel, in healthy volunteers.

Vaccines strategies: 70 volunteers will receive 3 DNA-C vaccinations and 1 NYVAC-C vaccination; 70 volunteers will receive 2 DNA-C vaccinations and 2 NYVAC-C vaccination.

DNA-C: 2x2ml intra muscular in right and left vastus lateralis; NYVAC-C: 1 ml intramuscular in non-dominant deltoid.

Main outcome:

1. the presence of CD8/CD4+ T cell responses defined according to internationally agreed criteria for evaluation of IFNgamma ELISPOT assays:

   * in response to env plus at least one of the gag, pol, nef peptide pools,
   * at weeks 26 or 28;
2. the safety parameters.

Secondary outcomes:

* cellular responses,
* antibody responses,
* all grade 1 and 2 adverse events,
* all events including those considered unrelated.

Sample size: 140 volunteers

Enrollment period: 9 months

Patient's participation duration: 78 weeks

Study duration: 27 months

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 55 years on the day of screening
* available for follow-up for the duration of the study (78 weeks from screening)
* able to give written informed consent
* at low risk of HIV and willing to remain so for the duration of the study low risk of HIV infection defined as:

  * no history of injecting drug use in the previous ten years
  * no gonorrhoea or syphilis in the last six months
  * no high risk partner (e.g. injecting drug use, HIV positive partner) either currently or within the past six months
  * no unprotected anal intercourse in the last six months, outside a relationship with a regular partner known to be HIV negative
  * no unprotected vaginal intercourse in the last six months outside a relationship with a regular known/presumed HIV negative partner
* willing to undergo a HIV test
* willing to undergo a genital infection screen
* if heterosexually active female, using an effective method of contraception with partner (combined oral contraceptive pill; injectable contraceptive; IUCD; consistent record with condoms if using these; physiological or anatomical sterility in self or partner) from 14 days prior to the first vaccination until 4 months after the last, and willing to undergo urine pregnancy tests prior to each vaccination
* if heterosexually active male, using an effective method of contraception with their partner from the first day of vaccination until 4 months after the last vaccination
* for French volunteers only :

  * subjects registered in French Health ministry computerised file and authorised to participate in a clinical trial
  * subjects covered by Health Insurance
  * subjects included in the ANRS vaccine research network of volunteers

Exclusion Criteria:

* pregnant or lactating
* clinically relevant abnormality on history or examination including history of grand-mal epilepsy; severe eczema; allergy to eggs or gentamicin; severe allergic diseases; liver disease with inadequate hepatic function; haematological, metabolic or gastrointestinal disorders; uncontrolled infection; autoimmune disease, immunodeficiency or use of immunosuppressives in preceding 3 months
* receipt of live attenuated vaccine within 60 days or other vaccine within 14 days of enrolment
* receipt of blood products or immunoglobin within 4 months of screening
* participation in another trial of a medicinal product, completed less than 30 days prior to enrolment
* history of severe local or general reaction to vaccination defined as

  * local: extensive, indurated redness and swelling involving most of the anterolateral thigh or the major circumference of the arm, not resolving within 72 hours
  * general: fever >= 39.5oC within 48 hours; anaphylaxis; bronchospasm; laryngeal oedema; collapse; convulsions or encephalopathy within 72 hours
* HIV 1/2 positive or indeterminate on screening
* positive for hepatitis B surface antigen, hepatitis C antibody or serology indicating active syphilis requiring treatment
* positive for DNA/ANA antibodies at titre considered clinically relevant by immunology laboratory
* grade 1 or above routine laboratory parameters (see section 4.1.4 & appendix 4 for definitions) Note of clarification 18th april 2008: hyperbilirubinemia has to be considered as an exclusion criterion only when confirmed to be conjugated bilirubinemia
* unlikely to comply with protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Immunogenicity parameter: presence of CD8/CD4+ T cell responses defined according to internationally agreed criteria for evaluation of IFNgamma ELISPOT assays, in response to env plus at least one of the gag, pol, nef peptide pools | week 26 and week 28
Safety parameter: grade 3 or above local adverse event, grade 3 or above systemic adverse event, grade 3 or above other clinical or laboratory adverse event,any event attributable to vaccine leading to discontinuation of the immunisation regimen. | within 72 weeks

SECONDARY OUTCOMES:
Cellular responses: CD8/CD4+ T cell mean IFNgamma Spot Forming Units (SFU) per million cells across the peptide pools | at weeks 26 and 28
Cellular responses: CD8/CD4+ T cell mean Spot Forming Units (SFU) per million cells across the peptide pools | at any week following the first immunisation including weeks 48 and 72
Cellular responses: mean proportion of CD4/CD8+ T cells producing IL-2 and/or IFNgamma following ex-vivo stimulation with HIV-1 peptide pools | at weeks 26 and 28, 48 and 72
Cellular responses: number of different epitopes that can be characterised | to be determined at a later stage
Antibody responses | to be determined at a later stage
All grade 1 and 2 adverse events | within 72 weeks
All events including those considered unrelated | within the 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yves LEVY, MD; PhD, Principal Investigator — Hôpital Henri Mondor-Créteil-France; Giuseppe PANTALEO, MD; PhD, Principal Investigator — Hospices CHUV-Lausanne-Switzerland
Locations (2):
- Hôpital Henri Mondor, Créteil, France
- Centre Hospitalier Universitaire Vaudois CHUV, Lausanne, Switzerland